CLINICAL TRIAL: NCT06250972
Title: Radiotherapy Plus Chemotherapy to Patients With CA19-9-elevated Advanced Pancreatic Cancer Who Are Not Refractory to Chemotherapy
Brief Title: Radiotherapy to Patients With CA19-9-elevated Advanced Pancreatic Cancer
Acronym: PTCA199-11
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-11
Record Dates: First submitted 2024-01-31; First posted 2024-02-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Irinotecan; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- chemotherapy (Active Comparator): Continuing chemotherapy using the previous regimen
  Interventions: Drug: Gemcitabine, Nab-paclitaxel, Irinotecan; Radiation: Intensity-Modulated Radiation Therapy (IMRT)
- Radiotherapy (Experimental): Patients will be recommended to receive Intensity-Modulated Radiation Therapy (IMRT) after about 2~6 cycles of chemotherapy. Other radiation therapies include stereotactic body radiotherapy (SBRT) and proton could be administered.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Drug: Gemcitabine, Nab-paclitaxel, Irinotecan — continuing chemotherapy using the previous regimen until disease progression
  Arms: chemotherapy
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Receive Intensity-Modulated Radiation Therapy (IMRT) after about 2~6 cycles of chemotherapy.

SUMMARY:
The purpose of this study is to evaluate the efficacy of chemotherapy plus radiotherapy to patients with CA19-9-elevated Advanced Pancreatic Cancer who are not refractory to chemotherapy.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. In 2011, the PRODIGE trial has shown that oxaliplatin, irinotecan, fluorouracil, and leucovorin (FOLFIRINOX) was associated with a survival advantage but had increased toxicity.

Carbohydrate antigen 19-9 (CA19-9) is the most widely used biomarker in pancreatic cancer. Circulating CA19-9 levels are positively correlated with tumor burden and stage in pancreatic cancer with a diagnostic sensitivity of approximately 80%, suggesting that approximately 20% of patients have normal CA19-9 levels. It is well recognized that Lewis (-) individuals, constituting approximately 10% of the population, have low or no secretion of CA19-9 due to the lack of critical enzyme involved in CA19-9 biosynthesis. Thus, approximately 10% of patients with pancreatic cancer have normal CA19-9 levels regardless of tumor stage. Our previously retrospective study has shown that CA19-9-normal advanced pancreatic cancer may be more sensitive to chemotherapy combined with radiotherapy.

The purpose of this study is to evaluate the efficacy of chemotherapy plus radiotherapy to patients with CA19-9-elevated Advanced Pancreatic Cancer who are not refractory to chemotherapy. Progression-free survival (PFS), objective response rate (ORR), overall survival (OS) and disease control rate (DCR) are measured every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed advanced pancreas adenocarcinoma.
* Patients who are not refractory to previous chemotherapy and who have not received radiotherapy.
* Locally advanced pancreatic cancer.
* Baseline serum CA19-9 > 37 U/mL, and CA19-9 level within normal range (≤37 U/mL) after chemotherapy .
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* The expected survival ≥ 3 months.
* Adequate organ performance based on laboratory blood tests.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Pregnant or nursing women.
* Primary pancreatic cancer.
* Baseline serum CA19-9 ≤ 37 U/mL.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
* Renal insufficiency or dialysis
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
* Patients who are allergic to oxaplatin or other chemotherapy drugs.
* Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival, PFS | At the end of Cycle 1 (each cycle is 28 days)
  PFS of subjects from recruiting to the time of disease progression

SECONDARY OUTCOMES:
Overall survival，OS | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from recruiting to the time of death from any cause
objective response rate (ORR) | At the end of Cycle 1 (each cycle is 28 days)
  CR + PR
disease control rate (DCR) | At the end of Cycle 1 (each cycle is 28 days)
  CR + PR + SD

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu X, Xiao Z, Liu H, Zhang P, Deng S, Ding L, Feng J, Luo J, Ni Q, Luo G, Yu X. Pancreatic Cancer: An Exocrine Tumor With Endocrine Characteristics. Ann Surg. 2024 Dec 1;280(6):e17-e25. doi: 10.1097/SLA.0000000000006168. Epub 2023 Dec 5. PMID 38050737
- [Background] Luo G, Jin K, Deng S, Cheng H, Fan Z, Gong Y, Qian Y, Huang Q, Ni Q, Liu C, Yu X. Roles of CA19-9 in pancreatic cancer: Biomarker, predictor and promoter. Biochim Biophys Acta Rev Cancer. 2021 Apr;1875(2):188409. doi: 10.1016/j.bbcan.2020.188409. Epub 2020 Aug 19. PMID 32827580
- [Background] Luo G, Liu C, Guo M, Long J, Liu Z, Xiao Z, Jin K, Cheng H, Lu Y, Ni Q, Yu X. CA19-9-Low&Lewis (+) pancreatic cancer: A unique subtype. Cancer Lett. 2017 Jan 28;385:46-50. doi: 10.1016/j.canlet.2016.10.046. Epub 2016 Nov 10. PMID 27840089